CLINICAL TRIAL: NCT01548443
Title: The Wound Healing Efficacy and Safety of Medifoam H in Patients With Minor, Acute Trauma: a Single-center, Randomized, Active-controlled, Open-label, Phase IV
Brief Title: Study to Evaluate Clinical Efficacy and Safety of "Medifoam H" in Wound Healing
Acronym: Medifoam H
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jong-Won Rhie, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP-MH-D01
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Trauma
Keywords: Wound Healing; hydrocolloid; Wound Dressing; Medifoam H; Duoderm THIN; Mild Acute Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medifoam H (Experimental): A group which treated with "medifoam H" on the wound.
  Interventions: Device: Medifoam H dressing
- Duoderm THIN (Active Comparator): A group which treated with " Duoderm THIN " on the wound
  Interventions: Device: Duoderm THIN dressing

INTERVENTIONS:
Device: Medifoam H dressing — Cover "medifoam H" on the wound for a week.
  Arms: Medifoam H
Device: Duoderm THIN dressing — Cover "Duoderm THIN" on the wound for a week
  Arms: Duoderm THIN

SUMMARY:
The wound healing efficacy and safety of "Medifoam H" in patients with minor, acute trauma.

The hypothesis of this study is that using "Medifoam H" dressing for a week is not inferior to using "Duoderm THIN" dressing in wound healing.

DETAILED DESCRIPTION:
This study is single-center, randomized, active-controlled, open-label, Phase IV to evaluate clinical efficacy of wound healing and safety of "Medifoam H" in patients with minor, acute trauma.

33 patients of treatment group and 33 patients of control group, total 66 patients will be enrolled to this study. Every patient will be treated with "Medifoam H" or "Duoderm THIN" for a week. During their participation, patients will visit 2 days and a week after to see investigator. Investigator will observe the wound and evaluate amount of exudation, infection status, wound healing.

ELIGIBILITY:
Inclusion Criteria:

1. Who has acute trauma(Laceration, Abrasion, Stitched wound, under superficial second-degree burn etc.)who satisfies at least 1 condition between followings:

1. Laceration, Stitched Wound: Length of under 10cm.
2. Abrasion, Burn: Total area of under 100㎠ , Depth of under 2mm. 2. Agreed to participate voluntarily in the study

Exclusion Criteria:

1. Who has hypersensitivity to hydrocolloid or its history.
2. Deep or severe infectious diseases of skin(example: Phlegmon, Abscess, Ulcer, Boil etc..) which is hard to treat with this investigational product.
3. A wound which is bitten by animal, human or inject. Or a wound has possibility of secondary infection through the tresis.
4. Who need surgical intervention for infection treatment.
5. Who has bacterial, viral, animal infectious disease
6. Who judged inappropriate to participate in the study by investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Wound healing rate according to amount of exudation at 1 week from baseline. If exudation is not existed, this will be defined as recovery | 0 to 1 week
  Wound healing rate according to amount of exudation at 1 week from baseline. If exudation is not existed, this will be defined as recovery. Exudation will be scored in 4 level: None/Mild/Normal/Severe.

SECONDARY OUTCOMES:
Rate of infection on wound | 1/3/7 days.
  Rate of infection on wound. Infection means pus, erythema or tenderness and this will be judged by observation of investigator and scored in 3 level: not present/minimally present/extensively present.
Amount of exudation at day 3. | 3 days
  Amount of exudation at day 3 from baseline. If exudation is not existed, this will be defined as recovery. Exudation will be scored in 4 level: None/Mild/Normal/Severe
Rate of wound healing | 3/7 days
  Rate of wound healing at day 3 and 7 from baseline. Would healing will be scored in 3 level: Better/Same/Worse.
Rate of changes in tissue after treatment | 3/7 days
  Rate of changes in tissue after treatment at day 3 and 7 from baseline. Changes in tissue will be recorded as percentage. Necrotic, sloughy, fibrous, granulation, epithelial, other tissues will be observed
Whether use of concomitant medication or not | 1/3/7 days
  Whether use of concomitant medication or not

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Won Rhie, MD.,PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, Seoul, South Korea